CLINICAL TRIAL: NCT07337811
Title: Selective Total Mesorectal Excision Based on Intra-Operative Frozen Section From Local Excision in Rectal Cancer Undergoing Neoadjuvant Chemoradiotherapy: A Prospective, Single-arm, Phase II Superiority Trial
Brief Title: Selective Total Mesorectal Excision Based on Intra-Operative Frozen Section From Local Excision in Rectal Cancer Undergoing Neoadjuvant Chemoradiotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Pei-Rong Ding, Director of the Department of Colorectal Surgery, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-FXY-237
Record Dates: First submitted 2025-07-27; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Rectal Cancer Patients
Keywords: Local Excision; Frozen Pathology; Chemoradiotherapy; Total Mesorectal Excision

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Selective Total Mesorectal Excision Based on Intra-Operative Frozen Section From Local Excision
  Interventions: Procedure: Selective Total Mesorectal Excision Based on Intra-Operative Frozen Section From Local Excision

INTERVENTIONS:
Procedure: Selective Total Mesorectal Excision Based on Intra-Operative Frozen Section From Local Excision — All participants undergo trans-anal full-thickness local excision under general anesthesia. The specimen is sent for intra-operative frozen-section pathology.
  ypT0-1 on frozen section → procedure concluded; patient enters watch-and-wait.
  ypT2-3 or R1 on frozen section → immediate completion total mesorectal excision (TME).
  Frozen-section ypT1-2 but final paraffin section up-staged to ypT2-3 or R1 → elective TME within 8 weeks.

SUMMARY:
This study is a prospective, single-arm, phase II superiority trial to determine whether a selective organ-preserving strategy based on immediate intra-operative frozen-section results can achieve favorable 2-year local control while lowering morbidity in patients with low rectal cancer (tumor ≤5 cm from the anus) who have a near clinical complete response (near-cCR) or partial response (residual tumor <2 cm) after radiation therapy.

Population: Adults with primary rectal adenocarcinoma located ≤5 cm from the anal verge who, after neoadjuvant radiotherapy, are judged to have near-cCR or partial response (residual tumor <2 cm).

Intervention: All participants undergo local excision under general anesthesia. The specimen is sent for intra-operative frozen section.

ypT0-1 on frozen section → procedure concluded; patient enters watch-and-wait. ypT2-3 or R1 on frozen section → immediate completion total mesorectal excision (TME).

Frozen-section ypT1-2 but final paraffin section up-staged to ypT2-3 or R1 → elective TME within 8 weeks.

Primary Endpoint: a composite outcome of 2-year local recurrence rate, surgical complications (≤30 days), and long-term functional impairment (anorectal, urogenital, and quality-of-life scales).

Secondary Endpoints: Agreement between intra-operative frozen-section pathology and final paraffin-section pathology, 3-year disease-free survival (DFS), 3-year overall survival (OS), surgery-sparing rate, post-operative recovery metrics, Quality-of-life scores.

Estimated Enrollment: 27 participants.

DETAILED DESCRIPTION:
Rectal cancer is a major global health burden with high morbidity and mortality. Its prognosis is generally worse than that of colon cancer, largely because of a higher risk of local recurrence. In 1982, Bill Heald introduced total mesorectal excision (TME), which has since proven to markedly reduce local recurrence. Peri-operative radiotherapy and chemotherapy further improve outcomes; pre-operative chemoradiotherapy (CRT) is superior to post-operative CRT, cutting local relapse by ~50%. Current National Comprehensive Cancer Network (NCCN) guidelines therefore recommend "pre-operative concurrent CRT followed by radical surgery" for locally advanced (stage II/III) rectal cancer. More recently, total neoadjuvant therapy (TNT) has refined this strategy, increasing pathologic complete response (pCR) rates to 20-40 %, and up to 60 % when combined with immunotherapy.

After neoadjuvant treatment, approximately 20 % of tumors achieve complete regression with pCR. If pre-operative assessment shows a clinical complete response (cCR), these patients may be offered an organ-preserving "watch-and-wait" approach instead of immediate TME, preserving sphincter function and quality of life. Since Habr-Gama's first report, multiple studies have confirmed the safety of this strategy: among patients managed by watch-and-wait, 15-20 % develop regrowth, 95 % of which are local and salvageable; 3-year distant-metastasis rates are only 8 % and 5-year cancer-specific survival is 94 %. Consequently, watch-and-wait is now standard for patients with cCR after CRT.

However, only 10-20 % of patients who ultimately achieve pCR are judged cCR pre-operatively. Imaging or endoscopic uncertainties (e.g., minimal ulceration) often lead to classification as partial response (PR) or near-cCR, depriving these patients of organ preservation. Traditionally, such patients proceed directly to TME. An emerging alternative is "local excision ± salvage TME": trans-anal full-thickness excision is performed first; if final pathology shows ypT0-1, no further surgery is required, whereas ypT2-3 or R1 margins trigger elective salvage TME. This risk-stratified approach aims to preserve organs in good responders while ensuring oncologic safety in poor responders.

Yet the GRECCAR-2 trial raised concerns: prior local excision may complicate subsequent TME, compromise sphincter preservation, and increase peri-operative morbidity (bleeding, infection, anorectal dysfunction) and long-term functional impairment. For patients with excellent tumor regression after CRT, these risks pose a dilemma.

To address this challenge, we propose the present clinical study, evaluating whether intra-operative frozen-section guidance during local excision can maintain diagnostic accuracy and oncologic safety while reducing the surgical complications and long-term functional sequelae associated with deferred TME.

This study is a prospective, single-arm, phase II superiority trial to determine whether a selective organ-preserving strategy based on immediate intra-operative frozen-section results can achieve favorable 2-year local control while lowering morbidity in patients with low rectal cancer (tumor ≤5 cm from the anus) who have a near clinical complete response (near-cCR) or partial response (residual tumor <2 cm) after radiation therapy.

Population: Adults with primary rectal adenocarcinoma located ≤5 cm from the anal verge who, after neoadjuvant radiotherapy, are judged to have near-cCR or partial response (residual tumor <2 cm).

Intervention: All participants undergo local excision under general anesthesia. The specimen is sent for intra-operative frozen section.

ypT0-1 on frozen section → procedure concluded; patient enters watch-and-wait. ypT2-3 or R1 on frozen section → immediate completion total mesorectal excision (TME).

Frozen-section ypT1-2 but final paraffin section up-staged to ypT2-3 or R1 → elective TME within 8 weeks.

Primary Endpoint: a composite outcome of 2-year local recurrence rate, surgical complications (≤30 days), and long-term functional impairment (anorectal, urogenital, and quality-of-life scales).

Secondary Endpoints: Agreement between intra-operative frozen-section pathology and final paraffin-section pathology, 3-year disease-free survival (DFS), 3-year overall survival (OS), surgery-sparing rate, post-operative recovery metrics, Quality-of-life scores.

Estimated Enrollment: 27 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed rectal adenocarcinoma.
2. Neoadjuvant therapy based on radiotherapy; post-radiotherapy evaluation ≥8 weeks later shows near clinical complete response (near-cCR) or partial response (PR) with residual tumor <2 cm.
3. Tumor distance from the anal verge ≤5 cm.
4. Age 18-75 years.
5. No synchronous multiple primary cancers.
6. No contraindications to pre-operative radiotherapy or chemotherapy.
7. Adequate organ function (cardiac, hepatic, renal, hematologic).
8. Patient or legally authorized representative able to understand the study protocol, willing to participate, and provide written informed consent.

Exclusion Criteria:

1. Age <18 or >75 years.
2. Concurrent or previous malignancy within the past 5 years (except adequately treated basal-cell or squamous-cell skin carcinoma or carcinoma in situ of the cervix).
3. Emergency surgery required for bowel obstruction, perforation, or bleeding.
4. Prior colorectal surgery that may compromise intestinal reconstruction.
5. Need for en-bloc multivisceral resection.
6. ASA physical status IV or V.
7. Pregnant or lactating women.
8. a) Women of child-bearing potential with a positive serum pregnancy test at baseline or who have not undergone pregnancy testing; post-menopausal women must have been amenorrheic for ≥12 months.
9. b) Men or women of reproductive potential unwilling to use effective contraception throughout the study period.
10. Severe psychiatric illness precluding informed consent or compliance.
11. Severe COPD, interstitial lung disease, or ischemic heart disease precluding safe surgery.
12. Continuous systemic corticosteroid therapy within 1 month before enrolment.
13. Contraindications to laparoscopic surgery.
14. Patient or legally authorized representative unable to understand the study conditions and objectives.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
2-year local recurrence rate | 2 years
  2-year local recurrence rate: defined as any clinical, radiologic, or pathologic evidence of tumor regrowth within the pelvis detected by digital rectal examination, endoscopy, CT/MR or PET-CT imaging, and biopsy (if indicated).
Rate of major surgical complications within 30 days post operation | 30 days
  Surgical complications graded ≥ III by the Clavien-Dindo classification (III = requiring surgical, endoscopic or radiologic intervention; IV = life-threatening complication requiring IC/ICU admission; V = death attributable to the complication).
Rate of permanent stoma at 2 years | 2 years
  Participants alive at 24 months who still have an end-colostomy or ileostomy deemed permanent by the treating surgeon.
Rate of anal incontinence at 2 years | 2 years
  Wexner score > 10 points assessed by validated questionnaire.
Rate of sexual dysfunction at 2 years | 2 years
  Sexual dysfunction assessed by the EORTC QLQ-C30/CR38 sexual function subscale; defined as score below reference value.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Rong Ding, Principal Investigator — Sun Yat-sen University
Locations (1):
- Dept. of Colorectal Surgery, Sun Yat-sen University Cancer Center. Yuexiu District, Dongfeng East Road 651, Guangzhou, Guanggong, China

IPD SHARING:
Plan to Share IPD: No